CLINICAL TRIAL: NCT03614546
Title: Clinical Trial of Radiotherapy in Treating Primary Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Department of oncology, Director of oncology department, The Third Xiangya Hospital of Central South University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-RT-002
Record Dates: First submitted 2018-07-15; First posted 2018-08-03 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Primary Hepatocellular Carcinoma
Keywords: primary hepatocellular carcinoma; radiotherapy; transarterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- A（surgery） group (Other): Hepatectomy
  Interventions: Procedure: Hepatectomy
- B1（SBRT） group (Experimental): Stereotactic Body Radiation Therapy(SBRT), 40-55Gy/5-6F
  Interventions: Radiation: SBRT
- B2a（TACE+ IMRT ） group (Experimental): First，treat with intensity modulated radiation therapy (IMRT),50Gy/25F/5W, 4 weeks after IMRT，treat with transcatheter arterial chemoembolization（TACE） 2-4 times
  Interventions: Radiation: IMRT; Procedure: TACE
- B2b（TACE+ IMRT ） group (Experimental): First，treat with transcatheter arterial chemoembolization（TACE） 2-4 times，4 weeks after TACE，treat with intensity modulated radiation therapy (IMRT),50Gy/25F/5W
  Interventions: Radiation: IMRT; Procedure: TACE
- C1（SBRT） group (Experimental): Stereotactic Body Radiation Therapy, 40-55Gy/5-6F
  Interventions: Radiation: SBRT
- C2a（TACE+ IMRT ） group (Experimental): First，treat with intensity modulated radiation therapy (IMRT),50Gy/25F/5W, 4 weeks after IMRT，treat with transcatheter arterial chemoembolization（TACE） 2-4 times
  Interventions: Radiation: IMRT; Procedure: TACE
- C2b（TACE+ IMRT ） group (Experimental): First，treat with transcatheter arterial chemoembolization（TACE） 2-4 times，4 weeks after TACE，treat with intensity modulated radiation therapy (IMRT),50Gy/25F/5W
  Interventions: Radiation: IMRT; Procedure: TACE

INTERVENTIONS:
Radiation: SBRT — Stereotactic Body Radiation Therapy (SBRT)
  Arms: B1（SBRT） group; C1（SBRT） group
Radiation: IMRT — Intensity-modulated Radiation Therapy (IMRT)
  Arms: B2a（TACE+ IMRT ） group; B2b（TACE+ IMRT ） group; C2a（TACE+ IMRT ） group; C2b（TACE+ IMRT ） group
Procedure: Hepatectomy — Hepatectomy
  Arms: A（surgery） group
Procedure: TACE — transarterial chemoembolization (TACE)
  Arms: B2a（TACE+ IMRT ） group; B2b（TACE+ IMRT ） group; C2a（TACE+ IMRT ） group; C2b（TACE+ IMRT ） group

SUMMARY:
The subjects of primary hepatocellular carcinoma diagnosed pathologically or clinically will be grouped according to the size, location, number and function of the liver, and respectively received Intensity-modulated Radiation Therapy (IMRT), Stereotactic Body Radiation Therapy (SBRT), Transarterial chemoembolization (TACE) or surgery.

DETAILED DESCRIPTION:
Primary hepatocellular carcinoma (HCC) is the sixth most malignant tumor in the world. In 2015, 466,000 people had been diagnosed as HCC in China, accounting more than half of the total incidence in the world; and 422,000 people died, making the HCC as the second reason for cancer related deaths in this country. Although many advances have been made in recent years in treatments such as Radiofrequency Ablation (RFA) and transarterial chemoembolization (TACE), the prognosis of patients with HCC is still poor. As a result, the prevention and treatments of HCC in China are still urgently needed to improve.

Being one of the three major treatments of cancer, radiotherapy has been used for HCC in very early times. In the pioneering days, however; whole-liver radiation was impossible to give lethal dose for cancer tissue due to the high risk of radiation induced liver disease (RILD) and even liver failure, which might lead to death of patients. Consequently, radiotherapy has long failed to play a major role in the treatment of liver cancer. But things are likely to be changed. In recent years, many research teams have applied precise external radiotherapy, such as intensity modulated radiation therapy (IMRT) and stereotactic body radiation therapy (SBRT), to the treatment of liver cancer, and has achieved good results. Despite of this, many guidelines still do not recommend radiotherapy as a first-line treatment for early and mid-term liver cancer due to the lack of high level of evidence from good clinical trials proving the effectiveness of SBRT/IMRT and other new radiotherapy techniques in the treatment of HCC.

In the investigator's previous clinical work, the investigators found that precise external radiotherapy such as SBRT and IMRT is effective in treating primary liver cancer. For example, patients with early stage HCC could achieve complete response (CR) after SBRT, and patients with local advanced HCC could be observed a significant reduction in the size of lesions and obvious improvement in the symptoms. Considering the poor prognosis of HCC and the shortcomings of surgery, RFA and TACE, the investigators then decided to carry out this multi-centered clinical trial of radiotherapy in HCC with the purpose of obtaining true and reliable clinical data and evidence, and focused on the following two questions: (1) whether radiotherapy, combined or not combined with TACE, could be a radical and first-line treatment for inoperable patients with early stage HCC; (2) what is the optimal sequence and timing of the combination of radiotherapy and TACE for patients with lesions adjacent to organs at risk and radical doses cannot be given. It is foreseeable that this clinical trial will change clinicians' understanding of the value of radiotherapy in the treatment of liver cancer, improve its status and even lead to revision of related guidelines/norms, and exert a far-reaching impact on the prognosis of patients with HCC.

The subjects who were pathologically or clinically diagnosed as primary liver cancer were grouped according to physical status, size/location/number of tumor, vascular invasion, extrahepatic metastasis, the relationship with organ at risk (OAR), and liver function. Then the subjects received IMRT, SBRT, TACE or surgery, and were followed up until the completion of treatment, the emergence of intolerance of toxicity, or the withdrawal of the trial.

Treatment methods:

1. Group A (surgery): surgical treatment (radical resection); 2. Group B (radiotherapy group 1):

1. Group B1 (SBRT): stereotactic radiotherapy (SBRT), 40-55Gy (Gray)/5-6F(Fractions), once daily.
2. Group B2a (IMRT+TACE): the subject firstly received IMRT, 50Gy/25F/5W (Weeks), once daily, and then TACE for 2-4 times at 4 weeks after radiotherapy.
3. Group B2b (TACE+IMRT): the subject firstly received TACE for 2-4 times, and then IMRT, 50Gy/25F/5W, once daily at 4 weeks after TACE.

3. Group C (radiotherapy group 2):

1. Group C1 (SBRT): stereotactic radiotherapy (SBRT), 40-55Gy/5-6F, once daily.
2. Group C2a (IMRT+TACE): the subject firstly received IMRT, 50Gy/25F/5W, once daily, and then TACE for 2-4 times at 4 weeks after radiotherapy.
3. Group C2b(TACE+IMRT): the subject firstly received TACE for 2-4 times, and then IMRT, 50Gy/25F/5W, once daily at 4 weeks after TACE.

During each scheduled visit in the treatment period, physical examination/weight, vital signs, hematology, coagulation, biochemistry, urine analysis, stool routine (occult blood) and other adverse events (AEs) and concomitant medication were evaluated.

Withdrawal Conditions:

1. subjects withdrew the informed consent;
2. treatment failure requiring additional emergency treatment (i.e. tumor progression or severe side effects caused by tumor emergencies);
3. AEs, if researchers and / or subjects hope or think it necessary to terminate treatment;
4. pregnancy;
5. Subject did not cooperate with the experimental treatment.
6. solid evidence of progression of the disease.

Termination conditions:

1. Evidence of ineffective treatment;
2. Security discovery preventing the continuation of the trial;
3. The applicant think that continuation of the trial is not in line with scientific or ethical principles.
4. The difficulty in the enrollment of subjects that makes it impossible for the completeness of the trial within an acceptable period of time.
5. The health authorities and the independent ethics committee (IECs) /institutional review board (IRBs) terminate the trial according to applicable regulations;
6. The health authorities require the suspension or termination of the trial.

Combined treatment

1. permissible treatment during the period of treatment; 1) Best supportive treatment; 2) Unconventional therapies including herbs or acupuncture and vitamins/ minerals; 3) Bisphosphonates can be used to treat bone metastases during treatment; 4) Active treatment for the combined diseases and all kinds of AE.
2. the prohibition of treatment during the treatment period 1) other local treatments for liver tumors including but not limited to any local ablation therapy or radioactive seed implantation; 2) systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnosis criteria of primary hepatocellular carcinoma: (1) primary hepatocellular carcinoma diagnosed by histology or cytology; (2) primary hepatocellular carcinoma diagnosed clinically (referring to the standard of diagnosis and treatment of primary hepatocellular carcinoma, version 2017);
2. Stage Ia-IIIa disease (referring to the standard of diagnosis and treatment of primary hepatocellular carcinoma, version 2017).
3. Child-Pugh score class A or B without encephalopathy;
4. Age between 18-80 years old;
5. At least one measurable lesion according to the 1.1 version of response evaluation criteria in solid tumors (RECIST).
6. ECOG(Eastern Cooperative Oncology Group) performance status of 0-2 at enrollment(subjects with ECOG performance status of 2 did not deteriorate in the last 2 weeks).
7. Written informed consent for the trial.
8. Be Willing and able to comply with planned visits, treatment plans, laboratory tests and other test procedures.
9. Have a life expectancy greater than 3 months judged by investigators；

Exclusion Criteria:

1. History of upper abdominal radiotherapy; 2. History of liver transplantation; 3. Abnormal laboratory results as follows:

1. abnormal hematology results, including hemoglobin less than 8.5 g/dL (no blood transfusion within 14 days before); neutrophils less than 1.5×109 /L or platelets less than 60×109 /L (no blood transfusion or growth factor was used within 7 days before);
2. abnormal liver function: total bilirubin >3×upper limit of normal (ULN); aspartate aminotransferase (AST) / alanine aminotransferase (ALT) > 5×ULN;
3. abnormal renal function: serum creatinine >1.5×ULN, or creatinine clearance rate (CrCl) < 60 mL/min according to Cockcroft-Gault formula.
4. international normalized ratio (INR) > 2.3 (according to the revised Child-Pugh grading Guide);
5. the calibration values of potassium, sodium, magnesium or calcium not within the normal range, and have clinical significance according to the judgment of the primary investigator.

4. History of other cancers besides primary hepatocellular carcinoma, with the exception of cured non-melanoma skin cancer, in situ cervical cancer, or other cancers received cured treatment and showed no signs of disease in at least 3 years.

5. Metastases to central nervous system (CNS) or brain; 6. Significant gastrointestinal bleeding occurred within 4 weeks before entering the trial.

7. Cardiac dysfunction as demonstrated by any of the following conditions:

1. recent echocardiography revealed a left ventricular ejection fraction < 45%.
2. severe arrhythmia;
3. unstable angina pectoris;
4. New York Heart Association III and IV congestive heart failure;
5. myocardial infarction occurred in the last 12 months before admission.
6. pericardial effusion; 8. Uncontrolled hypertension after standard treatment (blood pressure not stably below 150/90 mmHg) 9. Known human immunodeficiency virus (HIV) infection; 10. Pregnant or during lactation period, or is fertile male and female who is not willing or unable to take birth control/contraception to prevent pregnancy during the period between 2 weeks before radiation and 1 month after radiation; 11. Substance abuse, other acute or chronic physical or mental illness or abnormal laboratory examination that might increase the risk of participation judged by investigator.

12. Previous cancer treatment related toxicities that did not return to baseline or grade 0-1 (except for hair loss and peripheral neuropathy).

13. Any physical condition or illness that might increase the risk of participation judged by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to 5 years
  The time of patients from randomization to death caused by any cause.

SECONDARY OUTCOMES:
Disease control rate(DCR) | up to 5 years
  The proportion of patients who had a best response rating of complete response, partial response, or stable disease.
Progression free survival (PFS) | up to 5 years
  The time of patients from randomization to death caused by the progression of the tumor or any cause
Incidence of adverse events | up to 5 years
  Incidence of treatment-related adverse events assessed by CTCAE v4.0
Minimal volume of liver free from radiation | up to 5 years
  to explore the minimal volume of liver free from radiation in avoiding radiation-induced liver disease (RILD) during radiotherapy of primary hepatocellular carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: peiguo cao, doctor, Study Chair — The Third Xiangya Hospital, Central South University
Locations (1):
- The Third Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No